CLINICAL TRIAL: NCT06621147
Title: Application of Machine Learning Algorithms to Identify Optimal Candidates for Primary Tumor Resection in Patients with Metastatic Non-small Cell Neuroendocrine Tumors: Propensity Score Matching
Brief Title: Application of Machine Learning Algorithms to Identify Optimal Candidates for Primary Tumor Resection in Patients with Metastatic Non-small Cell Neuroendocrine Tumors
Acronym: MLA-MNSCLCNET
Status: Completed | Type: Observational
Sponsor: Hongquan Xing (Other)
Collaborators: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor-Investigator, Hongquan Xing, Doctor, Nanchang University
Organization: Nanchang University (Other)
Other Study IDs: NanchangU
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer - Non Small Cell
Keywords: lung cancer; machine learning; non-small cell neuroendocrine tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Demographic data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Surgery — Surgery

SUMMARY:
This study was based on public use data from the SEER database. The study did not require informed consent from the SEER registered cases, and the authors obtained Limited-Use Data Agreements from SEER.

DETAILED DESCRIPTION:
This study utilized publicly available data from the SEER (Surveillance, Epidemiology, and End Results) database, which is a comprehensive source of information on cancer statistics in the United States. The authors did not need to obtain informed consent from individuals whose cases are registered in the SEER database because the data is anonymized and is meant for public use. Instead, the authors acquired Limited-Use Data Agreements with SEER, which are legal contracts that allow researchers to access and use specific datasets under certain conditions while ensuring that the privacy of the individuals in the database is maintained. This agreement outlines the terms of data use, ensuring that the researchers adhere to guidelines for the ethical handling of data while still enabling them to conduct their research.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic Diagnosis of Non-Small Cell Neuroendocrine Carcinoma
* Known Surgical Information

Exclusion Criteria:

* Small cell lung cancer
* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with metastatic non-small cell neuroendocrine tumors
Sampling Method: Non-Probability Sample
Enrollment: 1776 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | The estimated time period for assessing events was January 2000 through December 2021. It is the time from random assignment to death from any cause (last follow-up for lost patients; end of follow-up for patients still alive at the end of the study).
  Overall survival refers to the duration of time from the start of diagnosis until death from any cause. It is a common endpoint used in clinical trials and medical research, particularly in oncology, to measure the effectiveness of a treatment or intervention. Overall survival provides a comprehensive picture of how well patients are doing and is often expressed as a percentage or a median time (e.g., the median overall survival time).